CLINICAL TRIAL: NCT01815723
Title: A Randomised, Double Blind, Double Dummy, Active Comparator and Placebo Controlled Confirmative Non-inferiority Trial of FP187 Compared to Fumaderm® in Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy Study on Dimethyl Fumarate to Treat Moderate to Severe Plaque Psoriasis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Forward-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP187-301; 2012-005685-35 (EudraCT Number)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Dimethyl fumarate; Fumaderm®
MeSH Terms: conditions — Psoriasis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- FP187 (Experimental): 500 mg FP187 daily (250 mg twice daily)
  Interventions: Drug: FP187; Drug: Fumaderm® placebo
- Dimethyl fumarate (Active Comparator): 720 mg Fumaderm® daily (240 mg three times daily)
  Interventions: Drug: Dimethyl fumarate; Drug: FP187 placebo
- Placebo (Placebo Comparator): Matching FP187 and Fumaderm® placebo
  Interventions: Drug: FP187 placebo; Drug: Fumaderm® placebo

INTERVENTIONS:
Drug: FP187 — 500 mg FP187 daily, two tablets of 125 mg twice daily, from 125 mg daily up-titrated to full dose over a 4-week phase, total treatment phase of 20 weeks
  Arms: FP187
Drug: Dimethyl fumarate — 720 mg Fumaderm® daily, two tablets of 120 mg three times daily, from 30 mg daily up-titrated to full dose over a 9-week phase, total treatment phase of 20 weeks
  Other Names: Fumaderm®
  Arms: Dimethyl fumarate
Drug: FP187 placebo — FP187 matching placebo tablets in the same regimen as for FP187 arm
  Arms: Dimethyl fumarate; Placebo
Drug: Fumaderm® placebo — Fumaderm® matching placebo tablets in the same regimen as for Fumaderm® arm
  Arms: FP187; Placebo

SUMMARY:
This multicenter, randomised, double-dummy, Fumaderm® and placebo-controlled, parallel-group study will compare the efficacy and safety of 500 mg of FP187 (250 mg twice daily) compared to 720 mg Fumaderm® (240 mg three times daily) over 20 weeks of treatment. After an initial wash-out non-drug treatment phase of 1 to 6 weeks, all patients will receive allocated Study treatment up-titrated to the relevant dose level (i.e., 500 mg daily FP187, 720 mg daily Fumaderm®, or placebo). The up-titration to full dose will last 4 weeks for FP187 and 9 weeks for Fumaderm®. After 20 weeks of treatment, all patients will be asked to enter a separate open label treatment protocol expected to continue for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* clinical diagnosis of stable moderate to severe plaque psoriasis for at least 6 months;
* clinical diagnosis of plaque psoriasis with an affected body surface area of no less than 10% and least 10 on the PASI scale and on the sPGA score at least as moderate;
* Besides psoriasis, patient is in good general health
* Patients with a DLQI score of at least 10

Exclusion Criteria:

* Pustular forms of psoriasis, erythrodermic or guttate psoriasis;
* Known immunosuppressive diseases;
* Presence of another serious or progressive disease including skin malignancies;
* Active skin disease;
* Use of topical medical treatment or UVB treatment during the 2 weeks preceding randomization;
* Use of systemic anti-psoriatic treatment preceding randomization: methotrexate, cyclosporine, steroids or PUVA (psoralen + UVA treatment) treatment within 4 weeks; biological treatment within 12 weeks; Stelara within 20 weeks; acitretin within 6 months;
* Treatment with Fumaderm® or other Dimethyl Fumarate containing products within 12 weeks prior randomization;
* Treatment with drugs influencing the course of psoriasis (e.g., antimalarial drugs, lithium) within 4 weeks prior to randomization;
* Treatment with retinoids, other immunosuppressive treatment, cytostatics or drugs with known harmful effects on the kidneys within 3 months prior to randomization;
* On-going stomach or intestinal problems;
* Aspartate transaminase (AST), Alanine transaminase (ALT) > 2 x upper normal limit (ULN), or Gamma-glutamyltransferase (γ-GT) > 2.5 x ULN;
* Creatinine Clearance < 60 ml/min;
* Leucopenia, eosinophilia or lymphopenia;
* Protein in the urine test;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a 75% reduction in their Psoriasis Area and Severity Index (PASI75) score from baseline | after 20 weeks of treatment
Responder rate of Static Physician's Global Assessment (sPGA) | after 20 weeks of treatment
  Achieving a score of clear or almost clear or a 2 step improvement on a 6-point scale as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kim A. Papp, MD, Principal Investigator — Probity Medical Research
Locations (1):
- Probity Medical Research, Waterloo, Ontario, Canada